CLINICAL TRIAL: NCT06135584
Title: Prospective Cohort Study on MAFLD-related Cirrhosis Prevention and Treatment Strategies
Brief Title: Study on MAFLD-related Cirrhosis Prevention and Treatment Strategies
Acronym: SMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Dysfunction-associated Fatty Liver Disease; Cirrhosis
Keywords: Treatment Strategies; Multicenter Real-World Study
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pioglitazone metformin tablets (Experimental): Pioglitazone metformin tablets 15mg/500mg (To control the fasting blood glucose below 7.0mmol/l, adjust the dose and dosage according to the blood glucose)
  Interventions: Drug: Pioglitazone metformin tablets
- Other drug (Active Comparator): Chinese patent medicine or Hypoglycemic drugs other than pioglitazone metformin tablets, pioglitazone, metformin and GLP1 ((To control the fasting blood glucose below 7.0mmol/l)
  Interventions: Drug: Other drugs
- Drug-free (Other): Drug-free
  Interventions: Other: Drug-free

INTERVENTIONS:
Drug: Pioglitazone metformin tablets — Drug intervention for 24 weeks and follow-up for another 72 weeks (fasting blood glucose was controlled below 7.0mmol/l throughout the study)
  Arms: Pioglitazone metformin tablets
Drug: Other drugs — Chinese patent medicine or hypoglycemic drugs other than pioglitazone metformin tablets, pioglitazone, metformin, GLP1
  Arms: Other drug
Other: Drug-free — Drug-free
  Arms: Drug-free

SUMMARY:
To establish a prospective, multicenter, biopsie-confirmed clinical cohort of MAFLD-related cirrhosis (F3-F4) in China, and analyze the clinical, histopathological features and natural outcomes of MAFLD-associated liver fibrosis/cirrhosis in China. And than to conducted a real-world study of different strategies of Chinese characteristics for the prevention and treatment of MAFLD-related cirrhosis to evaluate the efficacy and safety of the strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender and ethnicity are not limited;
2. Meet the diagnostic criteria for MAFLD;
3. F0-F4 stage of liver fibrosis confirmed by liver biopsy within 24 weeks;
4. Be willing to sign informed consent.

Exclusion Criteria:

1. Cirrhosis due to any chronic liver disease other than MAFLD (including but not limited to alcohol or drug abuse, medications, chronic hepatitis B or C, autoimmune, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency);
2. Any clinical evidence or history of peritonitis, varicose bleeding, or spontaneous encephalopathy;
3. According to the investigators' assessment, a history of heavy drinking for more than 3 months continuously within the previous year was selected. (Note: Heavy drinking was defined as more than 20 g per day on average for female subjects and more than 30 g per day for male subjects).
4. Use of NAFLD-related medication history (amiodarone, methotrexate, systemic glucocorticoids, tetracycline, tamoxifen, larger than hormone replacement doses of estrogen, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks within the year prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Controlled attenuation parameter (CAP) | Through study completion, an average of 96 week.
Transient elastography | Through study completion, an average of 96 week.
Model for end-stage liver disease score | Through study completion, an average of 96 week.
  Model for end-stage liver disease score ranges from 6 to 40 score (>40 calculated as 40 scores)，higher scores mean a worse outcome
Portalvein pressure gradient(HVPG) | Through study completion, an average of 96 week.
Prevalence of cirrhosis | Through study completion, an average of 96 week.
Prevalence of liver transplantation | Through study completion, an average of 96 week.
Prevalence of decompensated cirrhosis | Through study completion, an average of 96 week.

IPD SHARING:
Plan to Share IPD: No